CLINICAL TRIAL: NCT00052039
Title: A Randomized, Double-Blind, Three-Arm, Phase IIIb Study Comparing the Safety and Efficacy of Interferon Gamma-1b Alone, IFN-Gamma 1b With Azathioprine, and Azathioprine Alone in Patients With Idiopathic Pulmonary Fibrosis Receiving Prednisone
Brief Title: A Randomized, Double-Blind, Three-Arm, Phase 3b Study Comparing the Safety and Efficacy of Interferon Gamma-1b With Azathioprine, and Azathioprine Alone in Patients With IPF Receiving Prednisone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study design changes were needed based on GIPF-001 results
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIPF-003
Record Dates: First submitted 2003-01-21; First posted 2003-01-22 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Lung Disease; Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases; Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis | interventions — Interferon-gamma; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: interferon-gamma 1b — This study was terminated prior to enrollment.
Drug: azathioprine — This study was terminated prior to enrollment.

SUMMARY:
Study GIPF-003 is a Phase 3b study designed to define better therapeutic use of IFN-gamma 1b in patients wtih IPF. The study will be conducted primarily in Europe and will enroll 210 patients.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-04; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
This study was terminated prior to enrollment. | This study was terminated prior to enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Porter, MD, Study Director — InterMune
Locations (1):
- Ospedale S. Luigi Gonzaga - Regione, Torino, Orbassano, Italy